CLINICAL TRIAL: NCT03683992
Title: Early Outcomes of Cemented Versus Cementless Total Knee Arthroplasty Using the Triathlon Knee
Brief Title: Cemented vs Cementless TKA
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201308057
Record Dates: First submitted 2018-09-19; First posted 2018-09-25 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- cemented and cementless Triathlon group: cemented group are patients who get randomized to receive cemented knee implant and Patient randomized to receiving cement less knee implant.
  Interventions: Device: Triathlon total knee system

INTERVENTIONS:
Device: Triathlon total knee system — Implantable

SUMMARY:
The purpose of this study is to compare cemented and cementless versions of the Triathlon total knee arthroplasty/replacement (TKA) in terms of clinical outcomes, perioperative course, and outcome scores including function and patient satisfaction.

Patients who present to the clinical practices of Dr. Ryan Nunley, Dr. Robert Barrack, or Dr. Denis Nam and are suitable candidates for primary TKA will be screened for eligibility and invited to participate. Once enrolled participants will be randomized (1:1) to either receive a cemented or cementless Triathlon TKA. Data collected for the study will include standard of care clinical and radiographic evaluations collected during office visits and surgery, as well as study-specific patient questionnaires. Clinical, radiographic and questionnaire data will be collected pre-operatively, at the time of surgery, and at 6 weeks, 6 months, 1 year and beyond, and 2 years and beyond post-operatively. Patients will complete the following outcomes questionnaires preoperatively: New Knee Society Score, Oxford Knee Score, UCLA Activity Score, SF-12, and EQ-5D. The following questionnaires will be collected at four to six weeks, six months, one year and beyond, and two years and beyond postoperatively: New Knee Society Score, Forgotten Joint Score, Washington University Knee Satisfaction and Function Questionnaire, Oxford Knee Score, UCLA Activity Score, SF-12, and EQ-5D, and a Pain Drawing. In addition, a Pain Diary with a pain Visual Analog Scale (VAS) will be assessed once daily at home for 6 weeks after surgery.

DETAILED DESCRIPTION:
The purpose of this study is to compare cemented and cementless versions of the Triathlon total knee arthroplasty/replacement (TKA) in terms of clinical outcomes, perioperative course, and outcome scores including function and patient satisfaction.

Patients who present to the clinical practices of Dr. Ryan Nunley, Dr. Robert Barrack, or Dr. Denis Nam and are suitable candidates for primary TKA will be screened for eligibility and invited to participate. Once enrolled participants will be randomized (1:1) to either receive a cemented or cementless Triathlon TKA. Data collected for the study will include standard of care clinical and radiographic evaluations collected during office visits and surgery, as well as study-specific patient questionnaires. Clinical, radiographic and questionnaire data will be collected pre-operatively, at the time of surgery, and at 6 weeks, 6 months, 1 year and beyond, and 2 years and beyond post-operatively. Patients will complete the following outcomes questionnaires preoperatively: New Knee Society Score, Oxford Knee Score, UCLA Activity Score, SF-12, and EQ-5D. The following questionnaires will be collected at four to six weeks, six months, one year and beyond, and two years and beyond postoperatively: New Knee Society Score, Forgotten Joint Score, Washington University Knee Satisfaction and Function Questionnaire, Oxford Knee Score, UCLA Activity Score, SF-12, and EQ-5D, and a Pain Drawing. In addition, a Pain Diary with a pain Visual Analog Scale (VAS) will be assessed once daily at home for 6 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who qualify for a cementless primary total knee arthroplasty*
* 18 years of age but no more than 75 years of age
* Willing to be randomized
* Willing to sign informed consent
* Willing to return for all follow-up visits

Exclusion Criteria:

* Patients with inflammatory arthritis
* BMI equal to 40 or less.
* Patient with an active infection or suspected infection in the operative joint
* The absolute and relative contraindications stated in the FDA cleared labeling for the device
* Patients who have undergone osteotomy
* Patients who have had previous patella fracture or surgery
* Patients who have had previous healed tibia or femur fractures
* Patients who have had previous knee or hip replacement surgery on the ipsilateral side
* Patients who require patellar resurfacing
* Patients with major medical/muscular/orthopedic deformities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient between the ages of 18-75 getting a total knee surgery.
Sampling Method: Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Difference in tourniquet time | 1 year
  Tourniquet time will be recorded for each patient during surgery to see if there is a difference between tourniquet time between patients who are receiving cemented vs cementless.

SECONDARY OUTCOMES:
Difference in functional pain score | 2 years
  Patients will fill out a visual analog scale at 6 weeks, 1 year, 2 year to determine if there is a difference between functional pain score between cemented vs. cementless.
knee society score | 2 years
  Knee society score questionnaire will be completed preoperatively, 6 weeks, 1 year, and 2 year. Subscales are summed together to compute total score.
Forgotten joint score | 2 year
  Forgotten join score questionnaire will be completed preoperatively, 6 weeks, 1 year, and 2 year. Subscales are summed together to compute total score.
Oxford knee score | 2 years
  Oxford knee score questionnaire will be completed preoperatively, 6 weeks, 1 year, and 2 year.Subscales are summed together to compute total score.
UCLA Activity score | 2 year
  UCLA questionnaire will be completed preoperatively, 6 weeks, 1 year, and 2 year. Scale from 1 to 10. Higher number represent better outcome. Lower numbers represent worst outcome.
SF-12 questionnaire | 2 year
  SF-12 questionnaire will be completed preoperatively, 6 weeks, 1 year, and 2 year. Subscales are summed together to compute total score.
EQ-5D | 2 year
  EQ-5D questionnaire will be completed preoperatively, 6 weeks, 1 year, and 2 year. Subscales are summed together to compute total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University Medical School, St Louis, Missouri, United States